CLINICAL TRIAL: NCT07068841
Title: Study of the Pharmacokinetic Effect of Y-3 for Injection on Repaglinide Tablets, Warfarin Sodium Tablets, and Omeprazole Enteric-Coated Capsules in Healthy Participants
Brief Title: Pharmacokinetic Effect of Y-3 on Repaglinide，Warfarin and Omeprazole in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurodawn Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Y-3-LC-08
Record Dates: First submitted 2025-06-27; First posted 2025-07-16 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Pharmacokinetic Profiles; Y-3 for Injection; Drug-drug Interaction; Repaglinide Tablets; Warfarin Sodium Tablets; Omeprazole Enteric-coated Capsules; Safty
MeSH Terms: interventions — Warfarin; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- use of repaglinide, warfarin, and omeprazole or combined with Y-3 (Experimental)
  Interventions: Drug: sequentially single use of repaglinide, warfarin and omeprazole or combined with Y-3

INTERVENTIONS:
Drug: sequentially single use of repaglinide, warfarin and omeprazole or combined with Y-3 — Take repaglinide tablets, warfarin sodium tablets and omeprazole enteric-coated capsules without Y-3.
  Take repaglinide tablets, warfarin sodium tablets and omeprazole enteric-coated capsules sequentially during the use of Y-3.

SUMMARY:
The primary goal of this clinical trial is to evaluate the effect of Y-3 for injection on the pharmacokinetic profile of the sensitive finger substrates repaglinide tablets, warfarin sodium tablets, and omeprazole enteric-coated capsules for CYP2C8, CYP2C9, and CYP2C19 in Chinese healthy participants, to evaluate whether Y-3 for injection(40mg) will have clinical drug interactions with repaglinide tablets, warfarin sodium tablets and omeprazole enteric-coated capsules, so as to provide a reference for the drafting of Y-3 drug instructions for injection and a basis for the safe and rational use of the drug after marketing. The secondary goal of this clinical trial is to observe the effect of Y-3 for injection on the safety of repaglinide tablets, warfarin sodium tablets and omeprazole enteric-coated capsules. The main questions it aims to answer are:

* What the pharmacokinetic profiles of repaglinide tablets, warfarin sodium tablets, and omeprazole enteric-coated capsules when using Y-3 (40 mg) in healthy participants.
* If Y-3 for injection (40mg) will have clinical drug interactions with repaglinide tablets, warfarin sodium tablets and omeprazole enteric-coated capsules
* If Y-3 for injection (40mg) is safe in participants who using repaglinide tablets, warfarin sodium tablets, and omeprazole enteric-coated capsules.

Researchers will see what the pharmacokinetic profiles and safety of repaglinide tablets, warfarin sodium tablets, and omeprazole enteric-coated capsules when using Y-3 (40 mg) in healthy participants.

Participants will:

* Take repaglinide tablets, warfarin sodium tablets and omeprazole enteric-coated capsules without Y-3.
* Take repaglinide tablets, warfarin sodium tablets and omeprazole enteric-coated capsules during the use of Y-3.
* Answer questions regarding your medical history.
* Comply with the study procedures and requests.
* Complete all tests and collections of PK Sampling.
* Must not have any special dietary requirements and be able to consume the food (low-fat) provided by Tranquil Clinical Research during your 4-night stay.
* Must avoid excessive (> 8 cups per day) caffeine consumption (i.e. coffee or tea) during your time in the study.
* Must not consume any food or beverage rich in grapefruit, papaya, or mango during your time in the study.
* Must not take any other medications, including traditional Chinese medicines and herbal medicines, during your time in the study.
* Must avoid sexual activity or use non-drug contraceptive measures (i.e. condoms) during your time in the study.
* Female participants must not become pregnant while in the study.
* Must not receive any vaccinations during your time in the study.
* Must not donate blood for purposes outside of study procedures during your time in the study.
* Must not drink alcohol during your time in the study.
* Must not smoke during your time in the study.
* Inform your Study Doctor if you no longer wish to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* 1) Participants fully understand the purpose, nature, methods and possible adverse reactions of the trial, voluntarily act as participants, and sign the informed consent form before the start of any study procedures; 2) Healthy male or female participants aged 18 ~ 50 years old (including 18 and 50 years old); 3) Male weight ≥ 50.0 kg, female weight ≥ 45.0 kg, body mass index [BMI = weight (kg)/ height (m)2]: 19.0-26.0 kg/m2, including 19.0 and 26.0 kg/m2; 4) The results of vital signs, physical examination, 12-lead electrocardiogram examination, abdominal B-ultrasound (liver, gallbladder, pancreas, spleen, kidney), chest X-ray and laboratory examination (blood routine, urine routine, blood biochemistry, coagulation function, four items before blood transfusion, fecal occult blood examination) are normal or judged by the investigator to be abnormal of no clinical significance; 5) Participants (including male participants) have no fertility plan and voluntarily take effective contraceptive measures (contraceptive measures other than contraceptive drugs during the trial) within 3 months after signing the informed consent form to dosing, and have no sperm donation and egg donation plans; 6) Able to communicate well with the investigator, and understand and comply with the requirements of the trial.

Exclusion Criteria:

* 1) People with allergies: allergies to medicines, food, pollen, etc., or those who have a history of allergy to repaglinide tablets, warfarin sodium tablets, omeprazole enteric-coated capsules, Y-3 for injection or any of components of above investigational products; 2) Those who have diseases or medical history that may affect drug absorption, distribution, metabolism, excretion or interpretation of safety data, or diseases or medical history that can reduce compliance, including but not limited to gastrointestinal, renal, hepatic, pulmonary, neurological, hematological, endocrine, tumor, immunologic, psychiatric or cardiovascular and cerebrovascular diseases (especially liver and kidney insufficiency, diabetes, hypoglycemia, bleeding tendency or cachexia, malignant hypertension, thrombocytopenia); 3) Those who have undergone surgery within 6 months before the first use of the investigational products, or have undergone surgery that will affect the absorption, distribution, metabolism, and excretion of the investigational products, or plan to undergo surgery during the trial; 4) Those who have a history of fainting needle and blood sickness, cannot tolerate venipuncture blood collection, cannot tolerate intravenous administration and/or have difficulty in blood collection; 5) Those who cannot comply with the uniform diet (such as special dietary requirements, intolerance to standard meals, etc.); 6) For patients with creatinine clearance <80 mL/min, creatinine clearance (mL/min) = [(140-age) × body weight (kg)]/[72×Scr(mg/dl)] or creatinine clearance (mL/min) = [(140-age) × body weight(kg)]/[0.818×Scr(μmol/L)], female study participants were × 0.85 according to the calculated results; 7) Those who have participated in or are participating in other clinical trials within 3 months before the first use of the investigational products (drug clinical trial is defined as the use of clinical investigational products), or plan to participate in other clinical trials during the trial period or within 1 month after the end of the trial, or those who do not come to participate in clinical trials in person; 8) Those who have donated blood (including component blood) or had heavy bleeding (greater than 400 ml, except for blood loss during normal menstrual period in women) within 3 months before the first use of the investigational products, or received blood transfusion or used blood products, or plan to donate blood or blood components during the study or within 1 month after the end of the study; 9) Those who have had significant changes in diet or exercise habits within 3 months before the first use of the investigational products; 10) Those who have an average daily smoking volume of more than 5 cigarettes within 3 months before the first use of the investigational products, or cannot stop using any tobacco products (including any smoking cessation products containing nicotine) within 48 hours before the first use of the investigational products and during the trial; 11) Those who have a history of drug abuse or drug use within 6 months before the first use of the investigational products, or who are positive for drug abuse screening (morphine, methamphetamine, ketamine, tetrahydrocannabinolic acid, dimethylenedioxyamphetamine); 12) Those who have consumed more than 14 units of alcohol per week (1 unit of alcohol ≈ 360 mL of beer or 45 mL of spirits with 40% alcohol content or 150 mL of wine) per week within 3 months before the first use of the investigational products, or who cannot abstain from alcohol or stop using any diet containing alcohol within 48 hours before the first use of the investigational products and during the trial, or have a positive alcohol breath test result (greater than 0.0 mg/100 mL); 13) Those who consume excessive amounts of tea, coffee and/or caffeine-rich beverages (more than 8 cups, 1 cup = 250 mL) every day within 3 months before the first use of the investigational products, or cannot stop using caffeine-rich foods or beverages (such as chocolate, coffee, tea, cola, etc.) within 48 hours before the first use of the investigational products and during the trial; 14) Those who have used any drug that can change the activity of liver drug enzymes within 1 month before the first use of the investigational products; 15) Those who have been vaccinated within 1 month before the first use of the investigational products, or plan to receive any vaccine during the trial or within one week after the end of the trial; 16) Those who have used any prescription medicines, over-the-counter medicines, Chinese herbal medicines, health products and functional vitamins within 14 days before the first use of the investigational products; 17) Those who have one or more positive test results for hepatitis B surface antigen, hepatitis C virus antibody, HIV1/2 antigen/antibody and treponema pallidum antibody; 18) Females of childbearing potential who have had unprotected sex within 14 days prior to the first use of investigational products, or females who are pregnant or lactating, or who have a positive pregnancy test result; 19) Those who cannot stop ingesting grapefruit, dragon fruit, mango, lime, star fruit and other fruits or related products that affect metabolic enzymes within 48 hours before the first use of the investigational products and during the test; 20) Other conditions judged by the investigator to be inappropriate for enrollment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-05-18 (Actual); Primary Completion 2025-06-29 (Actual); Study Completion 2025-06-29 (Actual)

PRIMARY OUTCOMES:
Evaluate the AUC0-t of repaglinide in the healthy participants by venous blood and Phoenix WinNonlin. | on Day 1 and Day 16 of observation period
  Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration.
  Calculated according to linearity trapezoidal rule:
  AUC (i, i+1) = (Ti+1-Ti) (Ci+Ci+1) /2, and AUC0-t is the sum of all AUC (i, i + 1).
Evaluate the AUC0-t of S-warfarin in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration.
  Calculated according to linearity trapezoidal rule:
  AUC (i, i+1) = (Ti+1-Ti) (Ci+Ci+1) /2, and AUC0-t is the sum of all AUC (i, i + 1).
Evaluate the AUC0-t of omeprazole in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration.
  Calculated according to linearity trapezoidal rule:
  AUC (i, i+1) = (Ti+1-Ti) (Ci+Ci+1) /2, and AUC0-t is the sum of all AUC (i, i + 1).
Evaluate the AUC 0-∞of repaglinide in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 1, Day 16 of observation period.
  Area under the concentration-time curve from time 0 to infinity (extrapolated). AUC 0-∞ =AUC 0-t + Ct/λz (Ct is the last measured plasma concentration).
Evaluate the AUC0-∞ of S-warfarin in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Area under the concentration-time curve from time 0 to infinity (extrapolated). AUC 0-∞ =AUC 0-t + Ct/λz (Ct is the last measured plasma concentration).
Evaluate the AUC0-∞ of omeprazole in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Area under the concentration-time curve from time 0 to infinity (extrapolated). AUC 0-∞ =AUC 0-t + Ct/λz (Ct is the last measured plasma concentration).

SECONDARY OUTCOMES:
Evaluate the Cmax of repaglinide in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 1, Day 16 of observation period.
  Maximum observed plasma concentration. It was obtained directly from the measured plasma concentration-time data.
Evaluate the Cmax of S-warfarin in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Maximum observed plasma concentration. It was obtained directly from the measured plasma concentration-time data.
Evaluate the Cmax of omeprazole in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Maximum observed plasma concentration. It was obtained directly from the measured plasma concentration-time data.
Evaluate the Tmax of repaglinide in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 1, Day 16 of observation period.
  Time to reach maximum observed plasma concentration. It was obtained directly from the measured plasma concentration-time data.
Evaluate the Tmax of S-warfarin in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Time to reach maximum observed plasma concentration. It was obtained directly from the measured plasma concentration-time data.
Evaluate the Tmax of omeprazole in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Time to reach maximum observed plasma concentration. It was obtained directly from the measured plasma concentration-time data.
Evaluate the t1/2z of repaglinide in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 1, Day 16 of observation period.
  Terminal elimination half-life.
Evaluate the t1/2z of S-warfarin in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Terminal elimination half-life.
Evaluate the t1/2z of omeprazole in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Terminal elimination half-life.
Evaluate the λz of repaglinide in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 1, Day 16 of observation period.
  Terminal-phase elimination rate constant, slope of curves terminal segment at semi-log concentration-time curve calculated by linear regression.
Evaluate the λz of S-warfarin in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Terminal-phase elimination rate constant, slope of curves terminal segment at semi-log concentration-time curve calculated by linear regression.
Evaluate the λz of omeprazole in the healthy participants by venous blood and Phoenix WinNonlin. | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Terminal-phase elimination rate constant, slope of curves terminal segment at semi-log concentration-time curve calculated by linear regression.
Evaluate the AUC_%Extrap of repaglinide in the healthy participants by venous blood and Phoenix WinNonlin | On Day 1, Day 16 of observation period.
  The percentage of the AUC0-inf that has been extrapolated. AUC_%Extrap = [(AUC0-∞-AUC0-t)/AUC0-∞] × 100%
Evaluate the AUC_%Extrap of S-warfarin in the healthy participants by venous blood and Phoenix WinNonlin | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  The percentage of the AUC0-inf that has been extrapolated. AUC_%Extrap = [(AUC0-∞-AUC0-t)/AUC0-∞] × 100%
Evaluate the AUC_%Extrap of omeprazole in the healthy participants by venous blood and Phoenix WinNonlin | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  The percentage of the AUC0-inf that has been extrapolated. AUC_%Extrap = [(AUC0-∞-AUC0-t)/AUC0-∞] × 100%
Evaluate the Vz/F of repaglinide in the healthy participants by venous blood and Phoenix WinNonlin | On Day 1, Day 16 of observation period.
  Volume of distribution. Vz/F= CLz/F/λz
Evaluate the Vz/F of S-warfarin in the healthy participants by venous blood and Phoenix WinNonlin | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Volume of distribution. Vz/F= CLz/F/λz
Evaluate the Vz/F of omeprazole in the healthy participants by venous blood and Phoenix WinNonlin | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Volume of distribution. Vz/F= CLz/F/λz
Evaluate the CLz/F of repaglinide in the healthy participants by venous blood and Phoenix WinNonlin | On Day 1, Day 16 of observation period.
  Total body clearance. CLz/F=dosage/AUC0-∞
Evaluate the CLz/F of S-warfarin in the healthy participants by venous blood and Phoenix WinNonlin | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Total body clearance. CLz/F=dosage/AUC0-∞
Evaluate the CLz/F of omeprazole in the healthy participants by venous blood and Phoenix WinNonlin | On Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, Day 18, Day 19, Day 20, Day 22, Day 24 of observation period.
  Total body clearance. CLz/F=dosage/AUC0-∞
Evaluate the safety of repaglinide in the healthy participants taking Y-3 (40 mg) by the rate of adverse events. | Observation period and follow-up period. Day 1~Day 36.
  An AE is defined as any untoward medical event that occurs after receiving a drug or treatment or any deterioration of a disease or symptom that existed before receiving the investigational product or treatment (excluding the disease studied in this trial) in a subject or a clinical investigation subject, whether or not considered related to the investigational product or treatment. Therefore, an AE can be a discomfort sign (including an abnormal laboratory finding), symptom, or transient disease beyond any indication, whether or not related to the investigational product or treatment.
  The investigator will name each AE reported during the study by MedDRA PT and evaluate their severity using the criteria of "mild", "moderate" and "severe".
  The relevance evaluation is divided into 5 grades: 1-certainly related; 2- probably/likely related; 3-possibly related; 4-unlikely related; 5 not related.
Evaluate the safety of S-warfarin in the healthy participants taking Y-3 (40 mg) by the rate of adverse events. | Observation period and follow-up period. Day 1~Day 36.
  An AE is defined as any untoward medical event that occurs after receiving a drug or treatment or any deterioration of a disease or symptom that existed before receiving the investigational product or treatment (excluding the disease studied in this trial) in a subject or a clinical investigation subject, whether or not considered related to the investigational product or treatment. Therefore, an AE can be a discomfort sign (including an abnormal laboratory finding), symptom, or transient disease beyond any indication, whether or not related to the investigational product or treatment.
  The investigator will name each AE reported during the study by MedDRA PT and evaluate their severity using the criteria of "mild", "moderate" and "severe".
  The relevance evaluation is divided into 5 grades: 1-certainly related; 2- probably/likely related; 3-possibly related; 4-unlikely related; 5 not related.
Evaluate the safety of omeprazole in the healthy participants taking Y-3 (40 mg) by the rate of adverse events. | Observation period and follow-up period. Day 1~Day 36.
  An AE is defined as any untoward medical event that occurs after receiving a drug or treatment or any deterioration of a disease or symptom that existed before receiving the investigational product or treatment (excluding the disease studied in this trial) in a subject or a clinical investigation subject, whether or not considered related to the investigational product or treatment. Therefore, an AE can be a discomfort sign (including an abnormal laboratory finding), symptom, or transient disease beyond any indication, whether or not related to the investigational product or treatment.
  The investigator will name each AE reported during the study by MedDRA PT and evaluate their severity using the criteria of "mild", "moderate" and "severe".
  The relevance evaluation is divided into 5 grades: 1-certainly related; 2- probably/likely related; 3-possibly related; 4-unlikely related; 5 not related.
Evaluate the safety of repaglinide in the healthy participants taking Y-3 (40 mg) by the incidence of subject getting abnormal results of vital signs. | The whole study period. Day -14 ~ Day 36.
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Vital signs(blood pressure, respiration, pulse, body temperature） will be assessed by according equipments.(electronic sphygmomanometer，thermometer).
Evaluate the safety of S-warfarin in the healthy participants taking Y-3 (40 mg) by the incidence of subject getting abnormal results of vital signs. | The whole study period. Day -14 ~ Day 36
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Vital signs(blood pressure, respiration, pulse, body temperature） will be assessed by according equipments.(electronic sphygmomanometer，thermometer).
Evaluate the safety of omeprazole in the healthy participants taking Y-3 (40 mg) by the incidence of subject getting abnormal results of vital signs. | The whole study period. Day -14~Day 36.
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Vital signs(blood pressure, respiration, pulse, body temperature） will be assessed by according equipments.(electronic sphygmomanometer，thermometer).
Evaluate the safety of repaglinide in the healthy participants taking Y-3 (40 mg) by the incidence of subject getting abnormal results of physical examinations | The whole study period. Day -14 ~ Day 36.
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Physical examinations will be conduct by the investigator through observation.
Evaluate the safety of S-warfarin in the healthy participants taking Y-3 (40 mg) by the incidence of subject getting abnormal results of physical examinations | The whole study period. Day -14 ~ Day 36.
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Physical examinations will be conduct by the investigator through observation.
Evaluate the safety of omeprazole in the healthy participants taking Y-3 (40 mg) by the incidence of subject getting abnormal results of physical examinations | The whole study period. Day -14 ~ Day 36.
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Physical examinations will be conduct by the investigator through observation.
Evaluate the safety of repaglinide in the healthy participants taking Y-3 (40 mg) by the incidence of subject have infusion-related reactions | Observation period. Day 12~Day 25.
  infusion-related reactions is a general term for the adverse reactions related to infusion caused by the clinical use of intravenous preparations, including febrile reactions, circulatory overload reactions, phlebitis, air embolism, etc.
Evaluate the safety of S-warfarin in the healthy participants taking Y-3 (40 mg) by the incidence of subject have infusion-related reactions | Observation period. Day 12~Day 25.
  infusion-related reactions is a general term for the adverse reactions related to infusion caused by the clinical use of intravenous preparations, including febrile reactions, circulatory overload reactions, phlebitis, air embolism, etc.
Evaluate the safety of omeprazole in the healthy participants taking Y-3 (40 mg) by the incidence of subject have infusion-related reactions | Observation period. Day 12~Day 25.
  infusion-related reactions is a general term for the adverse reactions related to infusion caused by the clinical use of intravenous preparations, including febrile reactions, circulatory overload reactions, phlebitis, air embolism, etc.
Evaluate the safety of repaglinide in the healthy participants taking Y-3 (40 mg) by the incidence of subject getting abnormal results of laboratory tests | The whole study period. Day -14 ~ Day 36.
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Laboratory tests are composed of hematology, urinalysis, serum chemistry, coagulation test. Normal range is provided by the site.
Evaluate the safety of S-warfarin in the healthy participants taking Y-3 (40 mg) by the incidence of subject getting abnormal results of laboratory tests | The whole study period. Day -14 ~ Day 36.
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Laboratory tests are composed of hematology, urinalysis, serum chemistry, coagulation test. Normal range is provided by the site.
Evaluate the safety of omeprazole in the healthy participants taking Y-3 (40 mg) by the incidence of subject getting abnormal results of laboratory tests | The whole study period. Day -14 ~ Day 36.
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Laboratory tests are composed of hematology, urinalysis, serum chemistry, coagulation test. Normal range is provided by the site.
Evaluate the safety of repaglinide in the healthy participants taking Y-3 (40 mg) by the incidence of subject getting abnormal results of 12-lead ECG | The whole study period. Day -14 ~ Day 36.
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. 12-lead ECG will be analyzed by single RR Heart Rate, aggregate PR Interval, aggregate QRS Duration, aggregate RR Interval, aggregate QT Interval, aggregate QTC Interval. Normal range is provided by the site.
Evaluate the safety of S-warfarin in the healthy participants taking Y-3 (40 mg) by the incidence of subject getting abnormal results of 12-lead ECG | The whole study period. Day -14~Day 36.
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. 12-lead ECG will be analyzed by single RR Heart Rate, aggregate PR Interval, aggregate QRS Duration, aggregate RR Interval, aggregate QT Interval, aggregate QTC Interval. Normal range is provided by the site.
Evaluate the safety of omeprazole in the healthy participants taking Y-3 (40 mg) by the incidence of subject getting abnormal results of 12-lead ECG | The whole study period. Day -14 ~ Day 36.
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. 12-lead ECG will be analyzed by single RR Heart Rate, aggregate PR Interval, aggregate QRS Duration, aggregate RR Interval, aggregate QT Interval, aggregate QTC Interval. Normal range is provided by the site.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No